CLINICAL TRIAL: NCT02006875
Title: The Potential Benefit of 1-Hz rTMS to Improve Gross Motor Function After Stroke: A Randomized Controlled Trial.
Brief Title: rTMS Study to Improve Functional Performance for Patients With Stroke
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Principal Investigator, Yen-Nung Lin, Medical doctor of Department of Physical Medicine & Rehabilitation, Taipei Medical University WanFang Hospital
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 102-wf-eva-04
Record Dates: First submitted 2013-12-04; First posted 2013-12-10 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-12

CONDITIONS: Stroke
Keywords: repetitive transcranial magnetic stimulation; postural; balance; mobility; leg; stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- real rTMS (Experimental): Experimental included the a daily real rTMS session for 15 mins followed by a physical therapy for 45 mins.
  Interventions: Device: rTMS
- sham rTMS (Sham Comparator): the control interventions included a daily sham rTMS session for 15 minutes followed by a physical therapy for 45 minutes.
  Interventions: Device: rTMS

INTERVENTIONS:
Device: rTMS — Interventions started on the next weekday after pretest and were performed once a day for 15 consecutive weekdays. Participants in the E and C groups received rTMS (either real or sham, 1 Hz, 15 minutes), followed by a session of physical therapy for 45 minutes.
  Other Names: Magstim Rapid2

SUMMARY:
To use repetitive transcranial magnetic stimulation (rTMS) to treat stroke patients is getting a popular idea. Previous studies seemed to support its effects on facilitating motor recovery after stroke. This study focuses on the motor recovery of lower extremities. Investigators conducted the study to evaluate the treatment effect of rTMS on the functional performance of lower extremities in terms of postural control, balance, and mobility in stroke patients. Investigators hypothesized that these performances could be improved through the better motor control of lower extremities caused by rTMS.

DETAILED DESCRIPTION:
Protocol:

1. Setting: inpatient rehabilitation department of Shuang-Ho Hospital.
2. Study population: Patients received inpatient treatment or rehabilitation for stroke in Shuang-Ho Hospital (SHH).
3. Eligibility. Screening for eligibility was done by the 2 physiatrists from rehabilitation department of SHH.
4. Study design: controlled trial with stratified randomization
5. Blinding

   1. The patients were blinded by the real or sham coil of rTMS
   2. The assessors who performed the outcome measurements were blinded to the assignment of treatment.
6. Measurements.

   1. Baseline demographic records. The stroke severity was measured by National Institutes of Health Stroke Scale (NIHSS), Modified Rankin Scale (MRS), Brunnstrum stage, and Manual muscle test (MMT) before intervention.
   2. Clinical assessments.

      * Postural control was assessed by Postural Assessment Scale for Stroke Patients (PASS)
      * The motor recovery of lower extremities was assessed by the lower extremity subscale of Fugl-Meyer Assessment (FMA-LE)
      * The balance and gait subscales of Tinetti Performance Oriented Mobility Assessment (POMA-b and POMA-g)
      * Timed Up and Go (TUG) test was used to assess the gross mobility.
      * Barthel Index (BI) for the ADL independence
      * modified Rankin Scale (MRS) for disability classification were also collected.
   3. These measurements (including the clinical and corticomotor excitability assessments) are performed by one researcher who are responsible for the measurements.
7. Compliance and side effect. The compliance of interventions were investigated. The attendance of treatments (including rTMS sessions and physical therapy sessions) and possible side effect/discomfort were recorded during the interventions by a researcher. He also tries to understand the reason of drop-out from the study.

ELIGIBILITY:
Inclusion Criteria:

* unilateral hemiplegia caused by the stroke,
* first ever stroke,
* time since stroke: 10-90 days,
* age: 18-80 y/o,
* Functional ambulation classification (FAC): 0-2,

Exclusion Criteria:

* contraindication to TMS (eg, pacemaker, seizure history, pregnancy),
* cranial metal implants
* intracranial hemorrhage associated with tumor or arteriovenous malformation, craniotomy
* able to complete Timed Up and Go (TUG) test within 2 minutes
* unable to walk normally before the stroke
* those whose motor evoked potentials (MEP) of M1-UH were absent in the pretest

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Timed Up and Go (TUG) | Up to 3 months after interventions completed

SECONDARY OUTCOMES:
the lower extremity subscale of Fugl-Meyer Assessment (FMA-LE) | up to 3 months after the intervention completed
The balance and gait subscales of Tinetti Performance Oriented Mobility Assessment (POMA-b and POMA-g) | up to 3 months after the interventions completed
Barthel Index (BI) | Up to 3 months after interventions completed
Postural control was assessed by Postural Assessment Scale for Stroke (PASS) | up to 3 months after the intervention completed
  PASS which examines the patient's ability to maintain or change a given posture and is applicable to patients with very poor postural performance. This instrument has been reported to have a good validity and reliability at different recovery stages after stroke, minimal floor and ceiling effect, and be sensitive to changes in severe stroke patients at early stage after stroke.
modified Rankin Scale (MRS) | Up to 3 months after interventions completed

CONTACTS AND LOCATIONS:
Overall Officials: Yen-Nung Lin, MD, MS, Principal Investigator — Department of Physical Medicine and Rehabilitation, Wan Fang Hospital, Taipei Medical University
Locations (1):
- Shuang Ho Hospital, New Taipei City, Taiwan

REFERENCES:
- [Derived] Lin YN, Hu CJ, Chi JY, Lin LF, Yen TH, Lin YK, Liou TH. Effects of repetitive transcranial magnetic stimulation of the unaffected hemisphere leg motor area in patients with subacute stroke and substantial leg impairment: A pilot study. J Rehabil Med. 2015 Apr;47(4):305-10. doi: 10.2340/16501977-1943. PMID 25679340